CLINICAL TRIAL: NCT03895515
Title: The Effect of Fiasp® (Fast-acting Insulin Aspart) in Type 1 Diabetes Patients Using Continuous Glucose Monitoring / Flash Glucose Monitoring in Real-world Clinical Practice in Sweden. A Non-interventional, Retrospective Chart and Database Review Study
Brief Title: Effect of Fiasp® in Type 1 Diabetes Treatment
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN1218-4510; U1111-1228-4256 (Other: World Health Organisation (WHO))
Record Dates: First submitted 2019-03-27; First posted 2019-03-29 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Aspart

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fiasp®: Participants with type 1 diabetes who have switched to a basal-bolus insulin regimen with Fiasp® as the bolus insulin, from a basal-bolus insulin regimen with any other bolus insulin.
  Interventions: Drug: Fiasp®

INTERVENTIONS:
Drug: Fiasp® — Participants receive treatment with Fiasp® according to routine clinical practice. All treatment decisions, including assignment of participants to Fiasp® treatment, were made independently of the study and prior to the participants' inclusion in the study.

SUMMARY:
Fiasp® is a meal-time insulin that has been available in Sweden since June 2017. This study will investigate the effectiveness of Fiasp® in treating Type 1 Diabetes Mellitus. The study will be based on blood sugar measurements that the participants have uploaded to the Diasend® database and on existing data in their electronic medical records. The study does not require any additional visits to the study doctor.

ELIGIBILITY:
Inclusion criteria:

* Informed consent obtained before any study-related activities. Study-related activities are any procedures that are carried out as part of the study, including activities to determine suitability for the study (beyond identification of potential participants by searching for patients with type 1 Diabetes diagnosis, Fiasp® prescription information and electronic medical record (EMR) data to identify continuous glucose monitoring (CGM)/flash glucose monitoring (FGM) use
* Age greater than or equal to 18 years at the time of signing informed consent
* Switched to a basal-bolus insulin regimen with Fiasp® as the bolus insulin, from a basal-bolus insulin regimen with any other bolus insulin. Switch must have occurred greater than or equal to 26 weeks prior to data collection and during 01 September 2017 to 31 August 2018
* Treated with basal-bolus insulin regimen throughout the 26 weeks prior to Fiasp® initiation
* Treated with the same basal insulin, i.e. no records of switching the basal insulin, during the 26 weeks prior to Fiasp® initiation or the 26 weeks after Fiasp® initiation
* Diagnosed with type 1 diabetes for greater than or equal to 12 months prior to Fiasp® initiation
* Use of CGM/FGM during the 26 weeks prior to Fiasp® initiation and the 26 weeks after Fiasp® initiation
* Use of the same CGM/FGM device during the full 26-week period after Fiasp® initiation.

Exclusion criteria:

* Previous participation in this study. Participation is defined as signed informed consent
* Participation in clinical study with receipt of any investigational medicinal product known to affect glucose control during the 26-week period prior to Fiasp® initiation or the 26-week period after Fiasp® initiation
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation
* Patients prescribed any other glucose-lowering drugs than insulins (anatomical therapeutic chemical [ATC] class A10B), including oral and injectable drugs, as addition to their insulin treatment during the 26-week period prior to Fiasp® initiation or the 26-week period after Fiasp® initiation
* Use of Fiasp® as bolus insulin during the 26-week period prior to Fiasp® initiation
* Use of any insulin with an insulin pump (i.e. continuous subcutaneous insulin infusion) during the 26-week period prior to Fiasp® initiation or the 26-week period after Fiasp® initiation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with type 1 diabetes
Sampling Method: Non-Probability Sample
Enrollment: 178 (Actual)
Dates: Start 2020-01-03 (Actual); Primary Completion 2020-12-21 (Actual); Study Completion 2020-12-21 (Actual)

PRIMARY OUTCOMES:
Change in percentage of time spent in glycaemic target range (TIR) | Two-week period closest to and before index date, Two-week period closest to Week 26
  Measured in percentage point.
  The change in percentage of TIR was defined as a blood glucose level of 3.9 to 10.0 mmol/L after initiation of Fiasp® treatment. Index date is first Fiasp® prescription between 01 Sep 2017 and 01 Sep 2018.
  Time frame description:
  From: Closest continuous two-week period during the four weeks before the index date To: Continuous two-week period available closest to Week 26 during a period ranging between 20 weeks after index date to 32 weeks after index date. Measurements will, irrespective of analysis, only be considered if the patient is concomitantly on Fiasp® treatment.

SECONDARY OUTCOMES:
Change in mean sensor glucose | Two-week period closest to and before index date, Two-week period closest to Week 26
  Measured in mmol/L
  Index date is first Fiasp® prescription between 01 Sep 2017 and 01 Sep 2018.
  Time frame description:
  From: Closest continuous two-week period during the four weeks before the index date To: Continuous two-week period available closest to Week 26 during a period ranging between 20 weeks after index date to 32 weeks after index date. Measurements will, irrespective of analysis, only be considered if the patient is concomitantly on Fiasp® treatment.
Change in glycaemic variability (GV) (measured as coefficient of variation [CV]) | Two-week period closest to and before index date, Two-week period closest to Week 26
  Measured in percentage point
  Index date is first Fiasp® prescription between 01 Sep 2017 and 01 Sep 2018.
  Time frame description:
  From: Closest continuous two-week period during the four weeks before the index date To: Continuous two-week period available closest to Week 26 during a period ranging between 20 weeks after index date to 32 weeks after index date. Measurements will, irrespective of analysis, only be considered if the patient is concomitantly on Fiasp® treatment.
Change in percentage of time spent in level 1 hyperglycaemia (greater than 10.0 mmol/L) | Two-week period closest to and before index date, Two-week period closest to Week 26
  Measured in percentage point
  Index date is first Fiasp® prescription between 01 Sep 2017 and 01 Sep 2018.
  Time frame description:
  From: Closest continuous two-week period during the four weeks before the index date To: Continuous two-week period available closest to Week 26 during a period ranging between 20 weeks after index date to 32 weeks after index date. Measurements will, irrespective of analysis, only be considered if the patient is concomitantly on Fiasp® treatment.
Change in percentage of time spent in level 2 hyperglycaemia (greater than 13.9 mmol/L) | Two-week period closest to and before index date, Two-week period closest to Week 26
  Measured in percentage point
  Index date is first Fiasp® prescription between 01 Sep 2017 and 01 Sep 2018.
  Time frame description:
  From: Closest continuous two-week period during the four weeks before the index date To: Continuous two-week period available closest to Week 26 during a period ranging between 20 weeks after index date to 32 weeks after index date. Measurements will, irrespective of analysis, only be considered if the patient is concomitantly on Fiasp® treatment.
Change in percentage of time spent in level 2 hypoglycaemia (lesser than 3.0 mmol/L) | Two-week period closest to and before index date, Two-week period closest to Week 26
  Measured in percentage point
  Index date is first Fiasp® prescription between 01 Sep 2017 and 01 Sep 2018.
  Time frame description:
  From: Closest continuous two-week period during the four weeks before the index date To: Continuous two-week period available closest to Week 26 during a period ranging between 20 weeks after index date to 32 weeks after index date. Measurements will, irrespective of analysis, only be considered if the patient is concomitantly on Fiasp® treatment.
Change in percentage of time spent in level 1 hypoglycaemia (lesser than 3.9 mmol/L) | Two-week period closest to and before index date, Two-week period closest to Week 26
  Measured in percentage point
  Index date is first Fiasp® prescription between 01 Sep 2017 and 01 Sep 2018.
  Time frame description:
  From: Closest continuous two-week period during the four weeks before the index date To: Continuous two-week period available closest to Week 26 during a period ranging between 20 weeks after index date to 32 weeks after index date. Measurements will, irrespective of analysis, only be considered if the patient is concomitantly on Fiasp® treatment.
Proportion with CV lesser than 36% | Two-week period closest to Week 26
  Proportion of participants with/without GV corresponding to a CV lesser than 36%
  Time frame description:
  Continuous two-week period available closest to Week 26 during a period ranging between 20 weeks after index date to 32 weeks after index date. Measurements will, irrespective of analysis, only be considered if the patient is concomitantly on Fiasp® treatment.
Change in Glycated Haemoglobin A1c (HbA1c) | Latest measurement between Week -12 and index date, measurement closest to Week 26
  Measured in mmol/mol
  Index date is first Fiasp® prescription between 01 Sep 2017 and 01 Sep 2018.
  Measurement closest to Week 26 will be identified from a period ranging between 12 weeks after index date and 32 weeks after index date

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure 1452, Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Derived] Lind M, Catrina SB, Ekberg NR, Gerward S, Halasa T, Hellman J, Hess D, Londahl M, Qvist V, Bolinder J. Fast-Acting Insulin Aspart in Patients with Type 1 Diabetes in Real-World Clinical Practice: A Noninterventional, Retrospective Chart and Database Study. Diabetes Ther. 2023 Sep;14(9):1563-1575. doi: 10.1007/s13300-023-01444-y. Epub 2023 Jul 14. PMID 37450196